CLINICAL TRIAL: NCT00684593
Title: A Study to Assess the Clinical Effects of SCH 527123 in Psoriasis
Brief Title: A Study to Assess the Clinical Effects of Navarixin in Participants With Psoriasis (MK-7123-009)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P04481; 2006-006601-83 (EudraCT Number); P04481 (Other: Merck Protocol Number)
Record Dates: First submitted 2008-05-22; First posted 2008-05-26 (Estimated); Results first posted 2014-10-06 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2019-01

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis | interventions — navarixin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Navarixin (Experimental): Navarixin 30 mg administered orally once daily for 28 days.
  Interventions: Drug: Navarixin 10 mg
- Placebo (Placebo Comparator): Matching placebo to Navarixin administered orally once daily for 28 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Navarixin 10 mg — Navarixin capsules orally, once daily for 28 days.
  Arms: Navarixin
Other: Placebo — Matching placebo capsules to Navarixin orally, once daily for 28 days.
  Arms: Placebo

SUMMARY:
This study was conducted: 1) to assess the clinical effect of Navarixin on the Psoriasis Activity and Severity Index (PASI), 2) to determine the effects of Navarixin on the Physician's Global Assessment (PGA), 3) to evaluate the safety and tolerability of Navarixin, and 4) to determine the multiple-dose pharmacokinetics of Navarixin.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) 19 to 34, BMI = weight (kg)/height (m^2).
* Must have a diagnosis of psoriasis vulgaris (PASI >8) present for at least 1 year. Participants with an on-therapy PASI <=8 at Screening may be considered for inclusion. Participants must be discussed with the Sponsor prior to enrollment and the subject must have indicated that they are not satisfied with current therapy. To be included, participants must have a PASI >8 following washout of their current psoriasis therapy.
* Target lesion selected must be located on the head, trunk, arms or legs and be at least 10 cm^2 in size. The lesion's total numerical ratings for erythema, infiltration, and desquamation must be at least 6 out of the possible 12. Severity score for desquamation must be at least 2.
* Vital sign measurements (taken after ~3 minutes in a supine position) must be within the following ranges: oral body temperature between 35.0°C to 37.5°C; systolic blood pressure, 90 to 160 mm Hg; diastolic blood pressure, 45 to 90 mm Hg; pulse rate, 40 to 100 bpm.
* Have stable disease (ie, off treatment PASI during Screening period and Baseline PASI should not differ by more than 40%).
* Clinical laboratory tests (CBC, blood chemistries, and urinalysis) must be within normal limits or clinically acceptable to the investigator/sponsor. Participants must have a neutrophil count of at least 2 x 10^9/L to be included.
* Free of any clinically significant disease (other than psoriasis).
* Willing to give written informed consent and able to adhere to dose and visit schedules.
* For female participants: Negative serum pregnancy test (beta-hCG) and urine pregnancy test. Agree to use medically accepted methods of contraception during and for an appropriate pre-study period while receiving protocol specified medication, and for 1 month after stopping medication. Female participants of non-childbearing potential must be surgically sterilized or be postmenopausal.
* Male subject must agree to use an adequate form of contraception for the duration of the study.
* At Screening, ECG conduction intervals must be within gender specific normal range (ie, QTc for males <430 msec and females <450 msec) or if not within the normal range, the values must be considered clinically insignificant by the investigator and sponsor.

Exclusion Criteria:

* Female participants who are pregnant, intend to become pregnant (within 3 months of ending the study), or are breastfeeding.
* Participants who, in the opinion of the investigator, will not be able to participate optimally in the study.
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of any drug.
* History of any infectious disease within 4 weeks prior to drug administration and/or are positive for hepatitis B surface antigen, hepatitis C antibodies or human immunodeficiency virus (HIV).
* Immunocompromised participants.
* Positive screen for drugs with a high potential for abuse or have a history of drug or alcohol abuse in the past 2 years.
* History of mental instability or who have been treated for mood disorders.
* Donated blood in the past 60 days.
* Previous treatment with study medication.
* Currently participating in another clinical study or have participated in a clinical study within 30 days.
* Part of the study staff personnel or family members of the study staff personnel.
* Demonstrated clinically significant (requiring intervention) allergic reactions or who are known to be allergic to components of local anesthetics.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2007-06-01 (Actual); Primary Completion 2007-10-01 (Actual); Study Completion 2007-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=P04481&kw=7123-009&tab=access

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Navarixin | Placebo
Started | 21 | 10
Completed | 21 | 8
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Navarixin | Placebo | Total
Number analyzed (Participants) | 21 | 10 | 31
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.5 (10.5) | 43.9 (13.4) | 47.7 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 19 | 8 | 27

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change From Baseline in the Psoriasis and Activity Severity Index (PASI) Score at Day 29
Description: PASI score is a means to qualify the extent and severity of psoriatic lesions. The total score is calculated as the sum of the extent and severity of lesions on the head, arms, trunk, and legs and the score can range from 0 (no symptoms) to 72 (maximum symptoms).
Time Frame: Baseline and Day 29
Population: The population consisted of all treated participants with follow-up.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Groups:
- Placebo: Matching placebo to SCH 527123 administered orally once daily for 28 days.
Arm/Group | Navarixin | Placebo
Number analyzed (Participants) | 21 | 9
Score on a Scale | -3.30 (15.05) | -2.14 (13.26)

2. Secondary Outcome: Number of Participants by Physician's Assessment of Global Improvement (PGA) Score At Day 29
Description: The PGA is a questionnaire that asks the treating physician to rate the participant's signs and symptoms on a scale where 0=worse, 1=unchanged, 2= slight improvement, 3= fair improvement, 4= good improvement, 5= excellent improvement, and 6=cleared, with higher scores indicating better outcomes.
Time Frame: Day 29
Population: The population consisted of all treated participants with follow-up.
Measure: Number; unit: Participants
Arm/Group | Navarixin | Placebo
Number analyzed (Participants) | 21 | 9
Participants
  Score = 0 (worse) | 7 | 2
  Score = 1 (unchanged) | 6 | 2
  Score = 2 (slight improvement) | 8 | 4
  Score = 3 (fair improvement) | 0 | 1
  Score = 4 (good improvement) | 0 | 0
  Score = 5 (excellent improvement) | 0 | 0
  Score = 6 (cleared) | 0 | 0

3. Secondary Outcome: Mean Maximum Plasma Concentration (Cmax) of Navarixin at Day 28
Description: Participant blood samples were collected at 0, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, and 24 hours following oral administration of Navarixin to determine the mean Cmax at Day 28. Blood samples were not collected from the placebo group to evaluate this endpoint.
Time Frame: Day 28
Population: The population consisted of all participants for which serum samples were available for the determination of Cmax at Day 28. One participant was excluded due to erroneous blood sample collection relative to Navarixin dosing.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Navarixin
Number analyzed (Participants) | 20
ng/mL | 209.85 (51.50)

4. Secondary Outcome: Mean Area Under the Plasma Concentration-Time Curve From Time 0-24 Hours (AUC [0-24]) of Navarixin at Day 28
Description: Participant blood samples were collected at 0, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, and 24 hours following oral administration of Navarixin to determine the mean AUC(0-24) at Day 28. Blood samples were not collected from the placebo group to evaluate this endpoint.
Time Frame: Day 28
Population: The population consisted of all enrolled participants for which serum samples were evaluable at Day 28 for AUC (0-24). One participant was excluded due to erroneous blood sample collection relative to Navarixin dosing.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Navarixin
Number analyzed (Participants) | 20
hr*ng/mL | 420.37 (67.57)

5. Secondary Outcome: Mean Terminal Phase Half-life (T1/2) of Navarixin at Day 28
Description: Participant blood samples were collected at 0, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, and 24 hours to determine the mean T1/2 of Navarixin following oral administration at Day 28. Blood samples were not collected from the placebo group to evaluate this endpoint.
Time Frame: Day 28
Population: The population consisted of all enrolled participants for which serum samples were evaluable for T1/2. One participant was excluded due to erroneous blood sample collection relative to Navarixin dosing. An additional 2 participants were excluded from the population because their T1/2 was incalculable.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Navarixin
Number analyzed (Participants) | 18
Hours | 13.02 (6.63)

6. Secondary Outcome: Median Time to Maximum Plasma Concentration (Tmax) of Navarixin at Day 28
Description: Participant blood samples were collected at 0, 0.25, 0.5, 0.75, 1, 2, 3, 4, 6, 8, 10, 12, and 24 hours following oral administration of Navarixin to determine the Mean Tmax at Day 28. Blood samples were not collected from the placebo group to evaluate this endpoint.
Time Frame: Day 28
Population: The population consisted of all participants for which serum samples were available for the determination of Tmax at Day 28.
Measure: Median (Full Range); unit: Hours
Arm/Group | Navarixin
Number analyzed (Participants) | 21
Hours | 0.50 (51.50) [0.50 to 1.00]

ADVERSE EVENTS:
Time Frame: Up to Day 43
Arm/Group | Navarixin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/21 | 1/10
Other Adverse Events (participants affected / at risk) | 12/21 | 5/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Navarixin (N=21) | Placebo (N=10)
Venous Thrombosis Limb (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Navarixin (N=21) | Placebo (N=10)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 6 (6) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 5 (6) | 2 (5)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor shall have the right to review and comment with respect to publications, abstracts, slides, and manuscripts and the right to review and comment on the data analysis and presentation with regard to (1) proprietary information that is protected, (2) the accuracy of the information contained in the publication, and (3) to ensure that the presentation is fairly balanced and in compliance with FDA regulations.